CLINICAL TRIAL: NCT05988164
Title: "The Effect of Eye Masks Following Post-Gynecological Surgery on Sleep Quality: A Randomized Study"
Brief Title: "Eye Masks and Post-Surgical Sleep Quality"
Acronym: SEM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Dr. Kevser Ozdemir, Assosiated Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SAU-FHS-KI-02
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Sleep Quality
Keywords: Eye Mask; Sleep Quality; Gynecological Surgeries; Hospitalization; Health Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: There is an intervention group and a control group. Twenty-five participants participated in the intervention and 25 in the control group. Patients in the intervention group will be given eye masks and asked to sleep with them
Who Masked: Investigator
Masking Description: An independent statistician researcher, not directly involved in collecting patient data, will analyze the data to mask the investigator's influence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye mask Group (Experimental): Patients in the intervention group will be given eye masks and asked to sleep with them at 22:00 or earlier. Researchers or nurses will assist patients who cannot wear an eye mask at night. To measure patients' perception of sleep quality, we will use the Richard-Campbell Sleep Scale. The following morning, we will complete the post-test Richard-Campbell Sleep Scale to assess sleep quality.
  Interventions: Other: Eye Mask
- control Group (No Intervention): The control group will undergo no intervention, and their sleep quality will be measured in the hospital setting using the Richard-Campbell Sleep Scale.

INTERVENTIONS:
Other: Eye Mask — Patients in the intervention group will be given eye masks and asked to sleep with them at 22:00 or earlier.
  Arms: Eye mask Group

SUMMARY:
The aim of this study is to evaluate the impact of postoperative eye mask usage on sleep quality in patients who have undergone gynecological surgery.

DETAILED DESCRIPTION:
Sleep is considered a fundamental need for human health, and it contributes significantly to immune, mental, and physical functions. It has been shown that sleep quality influences individuals' quality of life, and it also promotes the healing process of injured tissues Sleep and rest are essential for optimal performance. In adults, 6-8 hours of sleep per day is required. Along with many unknown aspects of sleep's role in health and diseases, sleep deprivation is directly associated with poor mental and physical functions. In addition to compromising individuals' and public health, sleep deprivation can have severe complications for physical and behavioral functions.

Various factors contribute to sleep disturbances in the hospital environment. Sleep quality can be adversely affected by noise, light, and many other aspects of the surrounding environment. Non-pharmacological and pharmacological treatments can be used to improve sleep quality. Generally, non-invasive and cost-effective intervention methods are being used in hospitals to improve the quality of sleep during hospitalizing patients. Several studies have shown that using non-invasive tools like eye masks positively affects sleep quality. Nevertheless, there is no evidence that this tool is effective in patients undergoing gynecological surgery, and no studies have been founded locally to address this issue. Therefore, this study aims to examine sleep quality in women following gynecological surgery with eye masks.

Method:

A quasi-experimental design with a pre-test and post-test control group approach was used in this study. The quasi-experiment method uses a control group for experimental research. Two groups were randomly selected. There is an intervention group and a control group. Twenty-five participants participated in the intervention and 25 in the control group.

Patients in the intervention group will be given eye masks and asked to sleep with them at 22:00 or earlier. Researchers or nurses will assist patients who cannot wear an eye mask at night. The Richard-Campbell Sleep Scale will be used to measure patients' perceptions of sleep quality. The control group will undergo no intervention, and their sleep quality will be measured in the hospital setting using the Richard-Campbell Sleep Scale. Richards developed the Richard-Campbell Sleep Scale (RCSS) in 1987, and Karaman Zlü and Zer conducted its Turkish validity and reliability study in 2015. The scale consists of six items that evaluate the depth of nocturnal sleep, sleep onset latency, frequency of awakenings, duration of wakefulness after sleep onset, sleep quality, and noise level in the environment. Scale items are evaluated from 0 to 100 on a visual analog scale. Scores between "0-25" indicate very poor sleep, while scores between "76-100" indicate very good sleep. Participants' demographic characteristics, such as age, gender, narcotic drug consumption, average sleep duration before hospitalization, and sleep-facilitating tools, will be recorded on a participant information form developed in accordance with the literature. The post-test Richard-Campbell Sleep Scale will be used in the morning to assess sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Women who have undergone gynecological surgery Ability to read and speak Turkish participation with the ability to use an eye mask Patients who recovered at least six hours after surgery Patients with no traumatic or pathological head injury history Patients without sleep disorders or mental illnesses

Exclusion Criteria:

* Patients with an eye injury Patients who are allergic to eye masks Patients or their families who wish to withdraw from the study Patients with a mental or physical condition that makes participation in the study impossible.

Patients who cannot speak or read Turkish

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females aged 25-85 who underwent gynecological surgery are eligible to participate in this study..
Enrollment: 50 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-05-29 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Improving sleep quality with eye mask following gynecological surgery | 9 months
  Sleep quality and duration are increased in patients undergoing gynecological surgery with the use of postoperative eye masks. This results in reduced sleep interruptions and improved overall healthcare satisfaction and well-being of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
According to our ethics committee rules, there is no plan to make individual participant data (IPD) available to other researchers.